CLINICAL TRIAL: NCT06698679
Title: The Association Between Plasma Metabolites and the Risk, Efficacy and Prognosis in Early Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Caigang Liu, director of oncology, Shengjing Hospital
Other Study IDs: MUKDEN-METAB
Record Dates: First submitted 2024-11-13; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
Keywords: metabolites; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- cohort 1: women without breast cancer or other malignancies；breast cancer patients.
  Interventions: Other: No intervention
- cohort 2: patients diagnosed with breast cancer who received standard neoadjuvant therapy.
  Interventions: Other: No intervention
- Cohort 3: patients who have been discharged after breast cancer treatment.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There is no intervention in this study. We will obtain blood from the recruited patients and assess the metabolites therein. This is an observational work.

SUMMARY:
This study investigates plasma metabolites to clarify the relationship between these metabolites and breast cancer, aiming to identify valuable biomarkers. Furthermore, by incorporating clinical information-such as cancer stage, type, treatment outcomes, and prognosis-into prospective studies, the research seeks to further examine the correlation between plasma metabolites, treatment efficacy, and prognosis.

DETAILED DESCRIPTION:
Compared to normal tissues, tumor tissues exhibit significant metabolic changes. Consequently, tumor metabolic dysregulation is recognized as a novel marker of cancer. Differential analysis of metabolic phenotypes has the potential to establish new patient stratification criteria and biomarkers that facilitate personalized therapy. Breast cancer is the most prevalent malignant tumor among women. With advancements in metabolomics sequencing technology, an increasing number of researchers are focusing on the role of metabolomics in the diagnosis and treatment of breast cancer. It is important to note that the significance of individual metabolites in relation to breast cancer varies across studies; therefore, a standardized metabolic profile for assessing breast cancer risk has yet to be established.

This project collected data from natural populations and breast cancer patients by analyzing plasma metabolites alongside clinical treatment information. The goals of this study are to explore the correlation between plasma metabolites and breast cancer, as well as to identify biomarkers that characterize therapeutic efficacy and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1 Control Group: women without breast cancer or other malignancies. Case Group: patients with histologically confirmed carcinoma in situ or invasive breast cancer; no prior treatment; no distant metastasis; and not associated with other malignant tumor diseases.
* Cohort 2 Pathologically diagnosed as breast cancer; Treatment niave patients; To receive standard neoadjuvant therapy; Eastern Cooperative Oncology Group (ECOG) performance status of 0-1; Presence of at least one measurable lesion according to the Response Evaluation Criteria in Advanced Solid Tumors version 1.1 (RECIST v1.1) .
* Cohort 3 Patients who have been discharged after breast cancer treatment.

Exclusion Criteria:

* Histologically undiagnosed breast cancer. Breast cancer with distant metastases. Combined with other malignant tumors. Participants must not have participated in other clinical trials within the past month, unless those trials are observational or non-interventional in nature.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants included individuals without tumors, patients diagnosed with breast cancer , and patients who have been discharged after breast cancer treatment.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2031-06-30 (Estimated); Study Completion 2031-10-31 (Estimated)

PRIMARY OUTCOMES:
Cohort 1 : Different Plasma Metabolites | 2 years
  To measure the plasma metabolites of non-tumor individuals and breast cancer patients, and to analyze the differential metabolites between the two populations.
Cohort 2: Different Plasma Metabolites | 2 years
  pCR refers to the complete pathological remission of tumor lesions following neoadjuvant chemotherapy. To measure the plasma metabolites of breast cancer patients both before and after neoadjuvant chemotherapy, and to analyze the differential metabolites between patients who achieve pCR and those who do not.
Cohort 3: Different Plasma Metabolites | 7 years
  The metabolites in the blood of discharged breast cancer patients were measured regularly, and the differences in metabolites between patients with disease recurrence or metastasis and those without recurrence or metastasis within a 5-year period were analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No